CLINICAL TRIAL: NCT02223325
Title: Evaluation of Prognosis and Prognostic Scores in Geriatric Patients With Acute Pancreatitis: A Prospective Cohort Study
Brief Title: Evaluation of Prognosis and Prognostic Scores in Geriatric Patients With Acute Pancreatitis
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Gazi University (Other)
Responsible Party: Principal Investigator, Ibrahim Koral Onal, MD, associate professor, Gazi University
Other Study IDs: YOnal - 001
Record Dates: First submitted 2014-08-15; First posted 2014-08-22 (Estimated); Last update posted 2015-11-20 (Estimated); Status verified 2014-08

CONDITIONS: Acute Pancreatitis
Keywords: Elderly; Prognosis
MeSH Terms: conditions — Pancreatitis

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Elderly, acute pancreatitis: No intervention
- Adults <65 y, acute pancreatitis: No intervention

SUMMARY:
* To compare the prognosis of acute pancreatitis between geriatric and other adult patients
* To evaluate the efficacy of various prognostic scores in geriatric patients with acute pancreatitis

ELIGIBILITY:
Inclusion Criteria:

Acute pancreatitis Hospitalisation Adult patients

Exclusion Criteria:

* Recurrent pancreatitis
* Chronic pancreatitis
* Outpatient follow up
* Loss of follow up within 3 months of discharge

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Tertiary care patients
Sampling Method: Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2014-08; Primary Completion 2016-08 (Estimated)

PRIMARY OUTCOMES:
Mortality rate in geriatric patients with acute pancreatitis | Within 3 months

SECONDARY OUTCOMES:
Morbidity rate in geriatric patients with acute pancreatitis | Within 3 months

OTHER OUTCOMES:
The validity of various prognostic scores in geriatric patients with acute pancreatitis | Within 3 months